CLINICAL TRIAL: NCT04191538
Title: Conditioning Electrical Stimulation to Improve Outcomes in Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CES of CTS
Record Dates: First submitted 2019-12-03; First posted 2019-12-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Electrical Stimulation
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomized by an objective third party, who will provide electrical stimulation at the appropriate time given randomized cohort. Patients, surgeon, and investigator will be unaware of arm of study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conditioning electrical stimulation (Experimental): Patients will receive percutaneous electrical stimulation one week prior to carpal tunnel release. They will receive sham stimulation immediately after surgery to ensure blinding.
  Interventions: Procedure: Conditioning electrical stimulation
- Postoperative electrical stimulation (Active Comparator): Patients will receive electrical stimulation immediately following carpal tunnel release, per out previous studies. They will receive sham stimulation 1 week prior to surgery to ensure blinding.
  Interventions: Procedure: Postoperative electrical stimulation
- No electrical stimulation (Sham Comparator): Patients will not receive electrical stimulation. They will receive electrical stimulation before and after surgery to ensure blinding.
  Interventions: Procedure: No electrical stimulation

INTERVENTIONS:
Procedure: Conditioning electrical stimulation — Percutaneously, a small needle will be placed alongside the median nerve. Patients will receive 1 hour of 20Hz stimulation with voltage titrated to maintain patient comfort.
  Arms: Conditioning electrical stimulation
Procedure: Postoperative electrical stimulation — Immediately following carpal tunnel release, needles for electrical stimulation will be placed alongside the visualized median nerve. Patients will receive 1 hour of 20Hz stimulation with voltage titrated to maintain patient comfort.
  Arms: Postoperative electrical stimulation
Procedure: No electrical stimulation — Patients will receive sham stimulation (needles placed, no current delivered) pre- and post-operatively; however, no current will ever be delivered to the nerve. This is the control cohort.
  Arms: No electrical stimulation

SUMMARY:
Carpal tunnel syndrome is common, identified in 3% of the general population. Symptoms including numbness and pain are due to compression of the median nerve as it travels through a tunnel entering the wrist and can result in weakened grip strength and poor dexterity. Despite surgical release, nerve damage due to chronic compression often cannot be completely reversed, with resulting sensorimotor deficits. Postoperative electrical stimulation (ES) has been well-reported to improve nerve regeneration and is currently standard of practice at our institution. Investigators of this study have recently shown in an animal model that by changing the timing of the ES from postoperative to preoperative, this "conditioning" electrical stimulation (CES) significantly improves nerve regeneration.

Patients with severe carpal tunnel syndrome will be identified in plastic surgery clinics. Patients who consent to participating will undergo baseline testing including nerve conduction studies, sensory evaluation, motor testing, and patient-reported outcomes. Participants will be randomized to three groups: i) CES, ii) postoperative ES, and iii) no ES. CES will be delivered in clinic by placing a percutaneous needle alongside the median nerve, and stimulation will be delivered for one hour, with patient comfort dictating the voltage of stimulation. At the completion of one hour, the needle will be removed, and a standard carpal tunnel release will be performed by their plastic surgeon 4-7 days later. Patients will the second cohort will undergo postoperative ES immediately following their carpal tunnel release, using the same stimulation parameters as CES. The third cohort will receive only carpal tunnel release without stimulation.In all patients, sensory and motor reinnervation, using the same testing modalities as preoperative assessment, will be evaluated at 3, 6, and 12 months post-operative.

DETAILED DESCRIPTION:
Background: Carpal tunnel syndrome (CTS) is the most common compression neuropathy, with a population prevalence of 3%. One quarter of these patients have severe symptoms that necessitate surgical release. Our lab has previously demonstrated that electrical stimulation (ES) at 20Hz for 1 hour immediately following carpal tunnel release significantly improved terminal motor latency, sensory nerve conduction (1). Postoperative electrical stimulation enhances regeneration locally at the site of injury(2); by contrast, the conditioning lesion improves the rate of regeneration along the entire distal stump. The traditional conditioning lesion refers to a purposeful crush injury delivered to a nerve prior to its transection and repair. Despite 40 years of promising research at the bench, describing the conditioning lesion as an effective method of promoting regeneration and reinnervation in an animal model, translation to the bedside until recently has been impossible due to its injurious nature (3). Our laboratory has recently identified conditioning electrical stimulation (CES) as an effective method of enhancing axonal regeneration, and improve motor and sensory reinnervation (4). Investigators of this study have further shown that CES improves regeneration and sensorimotor reinnervation beyond that attainable by postoperative CES (unpublished data). As such preoperative CES is potentially a clinically feasible method of improving patient outcomes.

Hypothesis: ES delivered prior to carpal tunnel release will improve functional outcomes in patients with severe carpal tunnel syndrome.

Research Methods: Plastic surgeons in the Division of Plastic Surgeon will identify patients with severe carpal tunnel syndrome and obtain their consent to be considered for inclusion in this study. Inclusion criteria includes patients aged over 18 years who have failed conservative treatment, who are found to have severe carpal tunnel syndrome on nerve conduction studies (thenar motor unit loss minimum two standard deviations between the mean for the age group). Exclusion criteria includes patients with pre-existing peripheral neuropathies. Patients will be randomized to three treatment groups: a) CES, b) postoperative ES, and c) no ES. Carpal tunnel release will be performed by a plastic surgeon in the standard fashion without neurolysis of the median nerve.

In clinic, skin will be cleansed with alcohol and a small gauge needle will be placed percutaneously in the proximal forearm, along the course of the median nerve based on known surface anatomy. This needle will be connected to the cathode of an SD-9 Grass stimulator. The anode will be attached to an electrical cable placed more distally on the forearm. Stimulation protocol will be based on that traditionally used for postoperative ES: 20 Hz of continuous stimulation for one hour, with voltage titrated to maximize voltage without causing patient discomfort. At the completion of one hour, the needle will be removed. One week later, carpal tunnel release will be performed by the plastic surgeon per standard technique, without neurolysis of the median nerve. Among patients receiving postoperative ES, the cathode will be placed next to the median nerve proximal to the carpal tunnel at the time of surgical release, and electrical stimulation upon completion of the surgery will follow the same stimulation parameters as outlined for CES.

Primary outcomes include sensory testing (two-point discrimination, Semmes-Weinstein monofilament, and cold threshold), motor testing (Purdue Pegboard Test), and patient-reported outcomes (Disabilities of the Arm, Shoulder and Hand questionnaire). These are well established standard testing modalities for assessing recovery following carpal tunnel release (5). Scores for two-point discrimination range from 1 to 20 mm with smaller distance reflecting better hand sensibility. Mean score for the Purdue Pegboard Test in health control is 12 pegs with a greater number reflecting better hand dexterity. Range of score for the DASH questionnaire is 0 to 100 with a higher number representing greater disability. Testing will be performed preoperatively to establish baseline sensorimotor function, then postoperatively at 3, 6, and 12 months. Outcome measures will be analyzed using two-way ANOVA, with post-hoc analysis of significant association (p<0.05).

Justification: Recovery following surgical release in severe carpal tunnel is often incomplete, with persistent motor and sensory deficits. While postoperative ES improves regeneration, functional deficits persist; however, these studies have established ES as safe and well-tolerated by patients. By changing the timing of ES from postoperative to preoperative CES, animal data suggests functional outcomes can be further improved by upregulating regenerative pathways to maximize the rate of axonal extension. As CES can be delivered percutaneously in the clinic at the initial of initial assessment, prior to surgical release, this technique is both safe, clinically feasible and may significantly improve the outcomes of patients with compression neuropathies.

ELIGIBILITY:
Inclusion Criteria:

* Severe carpal tunnel syndrome (per screening nerve conduction test - thenar motor unit loss minimum two standard deviations between the mean for the age group)
* Failed conservative treatment (requires surgical intervention)

Exclusion Criteria:

* Preexisting neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Sensory reinnervation | Compare with baseline function to that at 12 months
  Patients will be tested for 2-point discrimination and touch (Semmes-Weinstein filaments)
Motor reinnervation | Compare with baseline function to that at 12 months
  Purdue Pegboard Test
Patient-reported outcome | Compare with baseline function to that at 12 months
  Disabilities of the Arm, Shoulder and Hand questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
All data collected will be de-identified and no individual information will be released.

REFERENCES:
- [Background] Gordon T, Amirjani N, Edwards DC, Chan KM. Brief post-surgical electrical stimulation accelerates axon regeneration and muscle reinnervation without affecting the functional measures in carpal tunnel syndrome patients. Exp Neurol. 2010 May;223(1):192-202. doi: 10.1016/j.expneurol.2009.09.020. Epub 2009 Oct 1. PMID 19800329
- [Background] Senger JLB, Verge VMK, Macandili HSJ, Olson JL, Chan KM, Webber CA. Electrical stimulation as a conditioning strategy for promoting and accelerating peripheral nerve regeneration. Exp Neurol. 2018 Apr;302:75-84. doi: 10.1016/j.expneurol.2017.12.013. Epub 2017 Dec 29. PMID 29291403